CLINICAL TRIAL: NCT01310946
Title: Establishment of Acute Lymphocytic Leukemia Data Base in the Department of Oncology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: RAC# 2021-051; RAC# 2021-051 (Other: KFSH&RC)
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: Acute Lymphocytic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Database Management Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Database — Database

SUMMARY:
Establishment of Acute Lymphocytic Leukemia Data Base in the Department of Oncology

DETAILED DESCRIPTION:
Establishment of Acute Lymphocytic Leukemia Data Base in the Department of Oncology

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed Acute Lymphocytic Leukemia

Exclusion Criteria:

* Patients with diagnosis other than Acute Lymphocytic Leukemia

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute Lymphocytic Leukemia Database
Sampling Method: Non-Probability Sample
Enrollment: 203 (Estimated)
Dates: Start 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: N Chaudhri, M.D., Principal Investigator — KFSH & RC
Locations (1):
- Kfsh & Rc, Riyadh, Saudi Arabia